CLINICAL TRIAL: NCT02833974
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, 8-week Treatment Study to Investigate the Safety, Pharmacodynamics, and Effect of the TLR7 Agonist, GSK2245035, on the Allergen-induced Asthmatic Response in Subjects With Mild Allergic Asthma
Brief Title: Effect of the GSK2245035 on the Allergen-induced Asthmatic Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205540; 2015-005645-31 (EudraCT Number)
Record Dates: First submitted 2016-07-12; First posted 2016-07-15 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-02

CONDITIONS: Asthma
Keywords: GSK2245035; TLR7 agonist; allergic asthma; FEV1
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2245035 20 ng (Experimental): Participants will receive 20 ng of GSK2245035 Nasal spray solution (1 spray=10 ng GSK2245035 per actuation per nostril) every week for the duration of 8 weeks administered using a metered Valois VP7 pump
  Interventions: Drug: GSK2245035 Nasal Spray Solution
- Placebo (Placebo Comparator): Participants will receive placebo Nasal spray solution (1 spray per nostril) every week for the duration of 8 weeks administered using a metered Valois VP7 pump
  Interventions: Drug: Placebo Nasal Spray Solution

INTERVENTIONS:
Drug: GSK2245035 Nasal Spray Solution — GSK2245035 Nasal Spray Solution 0.2 microgram (mcg)/mL delivering 10 ng GSK2245035 per actuation. A solution formulation in saline, preserved with Benzalkonium Chloride and Disodium Edetate.
  Arms: GSK2245035 20 ng
Drug: Placebo Nasal Spray Solution — Nasal Spray Solution as for GSK2245035 without active ingredient.
  Arms: Placebo

SUMMARY:
This study will assess whether Toll like receptor 7 (TLR7)-mediated pharmacology, with intranasal (i.n.) GSK2245035 20 nanogram (ng) administered weekly for a period of 8 weeks, will lead to reduced allergic reactivity in the lower airways in subjects with mild allergic asthma.

This will be a randomised, double-blind (sponsor open), placebo-controlled, parallel group, 8-week treatment study.

The study will consist of a screening period of up to approximately 4 weeks (involving two screening visits), a blinded treatment period of 8 weeks, followed by a follow-up period of up to 3 months. The total duration of the study for each subject will therefore be a maximum of approximately 6 months.

ELIGIBILITY:
Inclusion Criteria

* Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Diagnosis of asthma, as defined by the history of respiratory symptoms such as wheeze, shortness of breath, chest tightness and cough that vary over time and in intensity, together with variable expiratory airflow limitation for at least 6 months prior to screening
* Current asthma therapy. Intermittent short-acting beta-agonist (SABA) alone (on average for no more than 2 days per week)
* Positive skin prick test (3 mm or more greater than negative control) to common perennial or seasonal aeroallergen(s) (i.e., house dust mite, cat dander, grass pollen) at screening
* Pre-bronchodilator FEV1 > 70 % predicted normal at Screening Visit 1
* EAR with >=20 % FEV1 decrease between 5 and 30 minutes after the final allergen concentration is obtained at the screening bronchial allergen challenge (BAC) (decreases relative to the saline)
* LAR with three FEV1 decreases of >= 15 % between 4 and 10 hours after the final allergen concentration is obtained at the screening bronchial allergen challenge, with two FEV1 decreases being at consecutive time points (decreases relative to the saline)
* Subjects who are current non-smokers (defined as no use of any tobacco products in the 6-month period preceding the screening visit) and have a pack history of < 10 pack years. Number of pack years = (number of cigarettes per day/20) x number of years smoked
* Bodyweight >= 45kilograms (kg)
* Male OR female of non-reproductive potential Male subjects with female partners of child bearing potential complying with contraception requirements from the time of first dose of study medication until the final follow-up visit: Vasectomy with documentation of azoospermia, male condom plus partner use of one of the following contraceptive options: Contraceptive subdermal implant, Intrauterine device or intrauterine system, Oral contraceptive, either combined or progestogen alone, Injectable progestogen, Contraceptive vaginal ring, Percutaneous contraceptive patches. This is an all-inclusive list of those methods that meet the following GSK definition of highly effective: having a failure rate of less than 1% per year when used consistently and correctly and, when applicable, in accordance with the product label. For non-product methods (e.g., male sterility), the investigator determines what is consistent and correct use. The GSK definition is based on the definition provided by the International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH). The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception
* A female subject is eligible to participate if she is not pregnant, (as confirmed by a negative [serum or urine] human chorionic gonadotrophin [hCG] test), not lactating and where the following conditions applies: Non-reproductive potential: defined as pre-menopausal females with one of the following Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause [refer to laboratory reference ranges for confirmatory levels]). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment
* Capable of giving signed informed consent

Exclusion Criteria

* Alanine transaminase (ALT) >2xUpper Limit of Normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Heart rate corrected QT interval (QTc) > 450 milliseconds (msec) or QTc > 480 msec in subjects with Bundle Branch Block
* Asthma exacerbation requiring treatment with oral corticosteroids or hospitalization within 3 months prior to screening
* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures within the last 10 years
* Evidence of concurrent respiratory diseases such as pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, allergic bronchopulmonary aspergillosis, cystic fibrosis, bronchopulmonary dysplasia, or other respiratory abnormalities other than asthma
* Other concurrent diseases/abnormalities: A subject must not have any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study
* Respiratory tract infection that is not resolved within 2 weeks prior to screening
* Treatment with intranasal steroid, inhaled corticosteroid (ICS) with or without long-acting beta2-agonist (LABA), and treatment with non-ICS controller asthma medications (i.e., leukotriene modifier, methylxanthines) within 4 weeks prior to screening
* Use of long-acting antihistamines within 7 days' or short-acting antihistamines within 72 hours prior to the screening skin prick test
* Treatment with systemic corticosteroids within 6 weeks prior to screening
* Use of inhaled SABAs as rescue treatment on average for more than 2 days per week
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 units for males and females. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (~240 mililiter [ml]) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits
* Patient known to be intolerant to salbutamol or albuterol
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment
* A positive pre-study drug/alcohol screen
* A positive test for Human Immunodeficiency Virus (HIV) antibody
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Germany (4):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20762

REFERENCES:
- [Background] Siddall H, Quint D, Pandya H, Powley W, Shabbir S, Hohlfeld JM, Singh D, Lee L. Intranasal GSK2245035, a Toll-like receptor 7 agonist, does not attenuate the allergen-induced asthmatic response in a randomized, double-blind, placebo-controlled experimental medicine study. PLoS One. 2020 Nov 9;15(11):e0240964. doi: 10.1371/journal.pone.0240964. eCollection 2020. PMID 33166307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study investigated the safety, pharmacodynamics, and effect of the Toll-like receptor 7 (TLR7) agonist, GSK2245035, on allergen-induced asthmatic response in participants with mild allergic asthma. Participants received either intranasal 20 nanogram (ng) GSK2245035 or placebo once weekly for 8 weeks.
Pre-assignment Details: A total of 36 participants were randomized at different centers in United Kingdom and Germany..
Groups:
- Placebo: Participants received placebo matching GSK2245035 intranasal spray solution once weekly for 8 weeks
- GSK2245035 20 ng: Participants received 20 ng GSK2245035 intranasal spray solution at the rate of 1 spray per nostril (10 ng per actuation) once weekly for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | GSK2245035 20 ng
Started | 14 | 22
Completed | 13 | 19
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2245035 20 ng | Total
Number analyzed (Participants) | 14 | 22 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.6 (12.26) | 36.0 (11.65) | 36.3 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 12 | 21 | 33
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  African American/African Heritage | 0 | 2 | 2
  Asian - Central/South Asian Heritage | 0 | 1 | 1
  White | 14 | 19 | 33

OUTCOME MEASURES:

1. Primary Outcome: Late Asthmatic Response (LAR): Absolute Change From Saline in Minimum Forced Expiratory Volume in 1 Second (FEV1) Between 4-10 Hours Following Allergen Challenge One Week After Treatment
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to bronchial allergen challenge (BAC) at the one-week follow-up visit (one week after the eighth dose of the study treatment). Minimum FEV1 over 4-10 hours post-allergen challenge (minimum LAR) is the minimum value of all of the post-saline time points between 4 and 10 hours post-allergen challenge, inclusive of the 4 and 10 hours timepoints. Absolute change from saline in minimum FEV1 was calculated as the minimum FEV1 minus the saline FEV1 value. Per-Protocol Population comprises of all randomized participants who received at least one dose of study treatment and commence a BAC at follow-up and comply with the protocol.
Time Frame: Week 9
Population: Per-Protocol Population. Only those participants with data available at specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK2245035 20 ng
Number analyzed (Participants) | 10 | 17
Liters | -1.107 (0.7195) | -0.885 (0.5353)

2. Primary Outcome: LAR: Absolute Change From Saline in Weighted Mean FEV1 Between 4-10 Hours Following Allergen Challenge One Week After Treatment
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to BAC at the one-week follow-up visit (one week after the eighth dose of the study treatment). Weighted mean FEV1 over 4-10 hours post-allergen challenge includes all post-saline time points between 4 and 10 hours post-allergen challenge, inclusive of the 4 and 10 hours timepoints. The weighted mean FEV1 was derived by calculating the area under the curve, and dividing the value by the relevant time interval. Absolute change from saline at each time point was calculated as the highest allergen challenge FEV1 value minus the highest saline FEV1 value.
Time Frame: Week 9
Population: Per-Protocol Population. Only those participants with data available at specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK2245035 20 ng
Number analyzed (Participants) | 10 | 17
Liters | -0.546 (0.3932) | -0.576 (0.4018)

3. Secondary Outcome: Early Asthmatic Response (EAR): Absolute Change From Saline in Minimum FEV1 Between 0-2 Hours Following Allergen Challenge One Week After Treatment
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to BAC at the one-week follow-up visit (one week after the eighth dose of the study treatment). Minimum FEV1 over 0-2 hours post-allergen challenge (minimum LAR) is the minimum value of all of the post-saline time points between 0 and 2 hours post-allergen challenge, inclusive of the 0 and 2 hours timepoints. Absolute change from saline in minimum FEV1 was calculated as the minimum FEV1 minus the saline FEV1 value.
Time Frame: Week 9
Population: Per-Protocol Population. Only those participants with data available at specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK2245035 20 ng
Number analyzed (Participants) | 10 | 17
Liters | -1.246 (0.6052) | -1.096 (0.4113)

4. Secondary Outcome: EAR: Absolute Change From Saline in Weighted Mean FEV1 Between 0-2 Hours Following Allergen Challenge One Week After Treatment.
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to BAC at the one-week follow-up visit (one week after the eighth dose of the study treatment). Weighted mean FEV1 over 0-2 hours post-allergen challenge includes all post-saline time points between 0-2 hours post-allergen challenge, inclusive of 0 and 2 hours timepoints. The weighted mean FEV1 was derived by calculating the area under the curve, and dividing the value by the relevant time interval. Absolute change from saline at each time point was calculated as the highest allergen challenge FEV1 value minus the highest saline FEV1 value.
Time Frame: Week 9
Population: Per-Protocol Population. Only those participants with data available at specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK2245035 20 ng
Number analyzed (Participants) | 10 | 17
Liters | -0.604 (0.2670) | -0.587 (0.2388)

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinemia were categorized as SAE. Number of participants with AEs and SAEs have been reported.
Time Frame: Up to Week 20
Population: All Subjects Population comprise of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2245035 20 ng
Number analyzed (Participants) | 14 | 22
Participants
  Any AE | 10 | 21
  Any SAE | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormal Peak Expiratory Flow (PEF)
Description: The PEF is defined as the greatest rate of airflow that can be achieved during forced exhalation beginning with the lungs fully inflated. Participants were instructed to record their PEF readings each morning and evening into the diary card that was provided by the investigator. The minimum and maximum range ranges for PEF were <=205 and >=980 liters per minute.
Time Frame: Up to Week 12
Population: All Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2245035 20 ng
Number analyzed (Participants) | 14 | 22
Participants | 0 | 0

7. Secondary Outcome: Number of Participants Receiving Rescue Medication
Description: Salbutamol was administered as rescue medication only to participants who experienced serious discomfort. The data below exclude any Salbutamol administered as part of the planned study procedures (for example the Salbutamol administered after the Bronchial Allergen Challenge [BAC] is not counted as a rescue medication).
Time Frame: Up to Week 20
Population: All Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2245035 20 ng
Number analyzed (Participants) | 14 | 22
Participants | 1 | 2

8. Secondary Outcome: Number of Participants With Hematology Values of Potential Clinical Concern
Description: Blood samples were collected for analysis of hematology parameters. Hematology parameters included hematocrit, hemoglobin, platelet count, neutrophils, lymphocytes, monocytes, eosinophils, basophils, mean corpuscular volume, mean corpuscular hemoglobin, and red blood cells (RBC).
Time Frame: Up to Week 20
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2245035 20 ng
Number analyzed (Participants) | 14 | 22
Participants | 9 | 14

9. Secondary Outcome: Number of Participants With Clinical Chemistry Values of Potential Clinical Concern
Description: Blood samples were collected for analysis of clinical chemistry parameters. Clinical chemistry parameters included blood urea nitrogen, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, total protein, total and direct bilirubin, albumin, calcium, creatinine, glucose, potassium and sodium.
Time Frame: Up to Week 8
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2245035 20 ng
Number analyzed (Participants) | 14 | 22
Participants | 1 | 2

10. Secondary Outcome: Number of Participants With Abnormal Urine Analysis Findings
Description: Urine samples were collected for analysis of specific gravity, potential of hydrogen ions, glucose, protein, blood and ketones by dipstick method. Microscopic examination were performed if blood or protein values were abnormal.
Time Frame: Up to Week 8
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2245035 20 ng
Number analyzed (Participants) | 14 | 22
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events and non serious adverse events were collected from the start of study treatment up to Week 20
Description: All Subjects Population comprised of all participants who received at least one dose of study treatment.
Arm/Group | Placebo | GSK2245035 20 ng
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/22
Other Adverse Events (participants affected / at risk) | 10/14 | 21/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | GSK2245035 20 ng (N=22)
Headache (Nervous system disorders) | 8 | 9
Dizziness (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Parosmia (Nervous system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Rhinitis (Infections and infestations) | 1 | 1
Bacterial rhinitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Ear pruritus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1
Peak expiratory flow rate decreased (Investigations) | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT02833974/SAP_000.pdf
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT02833974/Prot_001.pdf